CLINICAL TRIAL: NCT00027066
Title: A Comparison of Warfarin and Aspirin for the Prevention of Recurrent Ischemic Stroke
Brief Title: Warfarin Versus Aspirin Recurrent Stroke Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Jay Preston Mohr, MD, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01NS028371 (NIH); R01NS028371 (NIH)
Record Dates: First submitted 2001-11-20; First posted 2001-11-21 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Stroke
Keywords: stroke; aspirin; warfarin
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Warfarin and Aspirin Placebo (Active Comparator): One 2 mg scored tablet daily of Warfarin and one 325 mg tablet daily of aspirin placebo.
  Interventions: Drug: Active Warfarin; Drug: Aspirin placebo
- Active Aspirin and Warfarin Placebo (Active Comparator): One 325 mg tablet daily of aspirin and one 2 mg scored tablet daily of Warfarin placebo.
  Interventions: Drug: Active Aspirin; Drug: Warfarin placebo

INTERVENTIONS:
Drug: Active Aspirin — 325mg tablet daily
  Arms: Active Aspirin and Warfarin Placebo
Drug: Active Warfarin — 2mg scored tablet daily
  Arms: Active Warfarin and Aspirin Placebo
Drug: Aspirin placebo — 325mg aspirin placebo pill
  Arms: Active Warfarin and Aspirin Placebo
Drug: Warfarin placebo — 2mg scored placebo tablet
  Arms: Active Aspirin and Warfarin Placebo

SUMMARY:
The goal of this study is to compare aspirin to warfarin for the prevention of recurrent stroke.

DETAILED DESCRIPTION:
This study compared aspirin to warfarin to determine optimal therapy for the prevention of recurrent stroke. Both drugs slow clotting of the blood. Blood clots are involved in the final stages of the most common type of stroke due to blockage of the vessels that supply oxygen-rich blood to the brain. Aspirin affects the blood platelets, while warfarin inhibits circulating clotting proteins in the blood. Numerous previous studies have proven that use of aspirin reduces recurrent stroke by about 25 percent. Part of the controversy about aspirin versus warfarin for stroke prevention has been the thinking among clinicians that warfarin may be a better blood thinner than aspirin to prevent almost all forms of stroke, but that it has greater side effects, increased risk of hemorrhage, and higher costs due to the need for blood tests to monitor the treatment effect for patients.

To make the aspirin and warfarin arms of the study as unbiased as possible, the investigators matched both groups of patients for primary stroke severity, age, gender, education, and race/ethnicity. The two groups were also matched for stroke risk factors, including hypertension, diabetes, cardiac disease, smoking, alcohol consumption, and physical activity. The investigators used an aspirin dose of 325 mg/day and a warfarin dose specifically tailored to each individual patient.

This study found that aspirin works as well as warfarin in helping to prevent recurrent strokes in most patients.

ELIGIBILITY:
Inclusion:

* Acceptable candidates for warfarin therapy
* Had an ischemic stroke within the previous 30 days
* Had scores of 3 or more on the Glasgow Outcome Scale

Exclusion:

* Base-line INR above the normal range (more than 1.4)
* History of stroke due to a procedure or that was attributed to high-grade carotid stenosis for which surgery was planned
* History of stroke associated with an inferred cardioembolic source

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2206
Dates: Start 1993-06; Primary Completion 2000-06 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. P. Mohr, M.D., Principal Investigator — Columbia University Health Sciences
Locations (1):
- Columbia University Health Sciences, New York, New York, United States